CLINICAL TRIAL: NCT03926949
Title: Outpatient Preoperative Parenteral Nutrition in Malnourished Surgical Patients: A Feasibility Study
Brief Title: Outpatient Preoperative Parenteral Nutrition in Malnourished Surgical Patients
Acronym: OPPortuNity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19G2208
Record Dates: First submitted 2019-04-15; First posted 2019-04-25 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Malnutrition; Surgery
MeSH Terms: conditions — Malnutrition | interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Participants will receive parenteral nutrition (Olimel 7.6% E 1000 ml), infused over 4-5 hours at outpatient infusion clinic for 5-10 days within 14 days prior to surgery.
  Interventions: Other: Parenteral Nutrition
- Control group (Other): Participants will receive nutrition therapy by registered dietitians within 14 days prior to surgery. Patients with SGA B and SGA C will receive advanced nutrition care and specialized nutrition care, respectively
  Interventions: Other: Standard Nutrition Care

INTERVENTIONS:
Other: Parenteral Nutrition — Olimel 7.6% E 1000 ml will be infused over 4-5 hours at outpatient infusion clinic for 5-10 days within 14 days prior to surgery.
  Other Names: Olimel 7.6% E 1000 ml
  Arms: Intervention group
Other: Standard Nutrition Care — Participants will receive nutrition therapy by registered dietitians within 14 days prior to surgery. Patients with SGA B and SGA C will receive advanced nutrition care and specialized nutrition care, respectively.
  Arms: Control group

SUMMARY:
Malnutrition is common in surgical patients. Many studies have shown a clear association between malnutrition and poor surgical outcomes. Parenteral nutrition (PN) is a nutrition intervention that is given by vein and can be safely provided to malnourished patients. It contains carbohydrates, fats, and protein just like you would normally in your diet. Pre-operative PN is able to improve outcomes in surgical patients. However, pre-operative PN has traditionally required hospital admission which results in increased length of stay, hospital cost, and hospital-acquired infection. Moreover, in hospital pre-operative PN may not be feasible or prioritized when access to inpatient surgery beds is limited. Outpatient PN provides the opportunity to solve this problem. The feasibility and impact of outpatient PN in malnourished patients undergoing major surgery have not previously been studied. This study aims to evaluate the feasibility of outpatient pre-operative PN and its effect on patient's outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Patients screened at risk of malnutrition by Canadian Nutrition Screening Tool (CNST) and identified as malnourished by subjective global assessment (SGA) B or C

Exclusion Criteria:

1. Patients undergoing minor or laparoscopic surgery
2. Pregnancy
3. Patients with severe systemic diseases defined by American Society of Anesthesiologists (ASA) classification III to V
4. Patients with diabetes mellitus
5. Patients with planned palliative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of parenteral nutrition completion | through study completion, an average of 1 year
  Rate of parenteral nutrition completion calculated by the number of patients who can complete parenteral nutrition before surgery for 5-10 days divided by total number of patients in parenteral nutrition group
Postoperative complications evaluated by Clavien-Dindo Classification | through study completion, an average of 1 year
  Clavien-Dindo Classification classifies postoperative complications into 5 grades (grade I to grade V) from mild to severe complications Grade I: no need specific intervention Grade II: need phamacological treatment Grade III: need surgical/endoscopic/radiological intervention Grade IV: life-threatening complications requiring ICU managment Grade V: death of a patient

SECONDARY OUTCOMES:
Length of hospital stay | through study completion, an average of 1 year
  Duration between hospital admission to discharge
Quality of life: Short Form (SF)-12 questionnaire | 5-10 days during parenteral nutrition infusion
  Quality of life evaluated by Short Form (SF)-12 questionnaire A mental component score (MCS-12) and a physical component score (PCS-12) are calculated by summation of mental and physical questions, respectively. The score range from 0-100, which the higher score means the better quality of life.
Body weight | 5-10 days during parenteral nutrition infusion
  Body weight measurement in kilograms
Nutrition status | 5-10 days during parenteral nutrition infusion
  Nutrition status evaluated by patient-generated subjective global assessment
  Patient-generated subjective global assessment divides a patient into 3 groups:
  A = well-nourished B = moderately malnourished or suspected malnutrition C = severely malnourished The total score is also calculated by summation of scores from weight, food intake, gastrointestinal symptoms, activity, metabolic demand, and physical examination. It ranges from 0-55, which the lower score means the better nutrition status.
Muscle power | 5-10 days during parenteral nutrition infusion
  Muscle power evaluated by handgrip strength test
Cost-saving | through study completion, an average of 1 year
  Difference in total length of stay (primary length of stay plus length of stay during readmission) between 2 groups multiplies by estimated unit cost of inpatient hospital stay per day from Alberta Health Service
Hospital readmission | 30 days after discharge
  Readmission rate within 30 days after discharge
Total energy from parenteral nutrition | 5-10 days during parenteral nutrition infusion
  Total energy from parenteral nutrition measured by total energy in kilocalories per day multiply by total days of parenteral nutrition
Total protein from parenteral nutrition | 5-10 days during parenteral nutrition infusion
  Total protein from parenteral nutrition measured by total protein in grams per day multiply by total days of parenteral nutrition
Acceptability, appropriateness, and feasibility of intervention measured by Acceptability, Appropriateness, and Feasibility Questionnaire | through study completion, an average of 1 year
  Acceptability, Appropriateness, and Feasibility Questionnaire included score 1 to 5
  1. completely disagree with intervention
  2. disagree with intervention
  3. neither agree nor disagree with intervention
  4. agree with intervention
  5. completely agree with intervention

CONTACTS AND LOCATIONS:
Overall Officials: Leah Gramlich, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Undecided